CLINICAL TRIAL: NCT01444742
Title: Clofarabine Plus Low-Dose Cytarabine for the Treatment of Patients With Higher-Risk Myelodysplastic Syndrome (MDS) Who Have Been Relapsing After, or Are Refractory to, Hypomethylator Therapy
Brief Title: Clofarabine Plus Low-Dose Cytarabine for Patients With Higher-Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0660; NCI-2011-03436 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-09-28; First posted 2011-10-03 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Leukemia; Myeloproliferative Diseases
Keywords: Leukemia; Myeloproliferative Diseases; Myelodysplastic Syndrome; (MDS); Relapsing; Refractory; Clofarabine; Clofarex; Clolar; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Recurrence | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Clofarabine + Cytarabine (Experimental): Induction:
  Clofarabine 10 mg/m2 1-2 hours by vein daily for 5 days (days 1-5) Cytarabine 20 mg subcutaneously twice daily for 7 days (days 1-7)
  Consolidation:
  Clofarabine 10 mg/m2 1-2 hours by vein daily for 3 days (days 1-3) Cytarabine 20 mg subcutaneously twice daily for 5 days (days 1-5)
  Interventions: Drug: Clofarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Clofarabine — Induction:
  10 mg/m2 by vein over 1-2 hours daily for 5 days (days 1-5)
  Consolidation:
  10 mg/m2 by vein over 1-2 hours daily for 3 days (days 1-3)
  Other Names: Clofarex; Clolar
Drug: Cytarabine — Induction:
  20 mg subcutaneously twice daily for 7 days (days 1-7)
  Consolidation:
  20 mg subcutaneously twice daily for 5 days (days 1-5)
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine Arabinosine Hydrochloride

SUMMARY:
The goal of this clinical research study is to learn if clofarabine when given in combination with cytarabine can help to control myelodysplastic syndrome (MDS) after the disease could not be controlled with standard therapy. The safety of this treatment will also be studied.

Clofarabine is designed to interfere with the growth and development of cancer cells.

Cytarabine is designed to insert itself into DNA (the genetic material of cells) of cancer cells and stop the DNA from repairing itself.

DETAILED DESCRIPTION:
Induction Cycles:

If you are found to be eligible to take part in the study, on Days 1-5 of each cycle , you will receive clofarabine by vein over 1-2 hours.

On Days 1-7 of each cycle, you will receive cytarabine by injection under the skin over several seconds 2 times a day.

You may receive up to 3 cycles at this dose and schedule (also called "induction cycles"). There are 7 treatment days in each cycle but the total length of one cycle (including rest and recovery period) is usually between 4 and 8 weeks.

Consolidation Cycles:

After you have completed the Induction Cycles, if you show a response to treatment, you can then continue with up to a total of 12 more cycles of therapy, which will be called "consolidation cycles". Not every participant may be able to receive all 12 consolidation cycles. The actual number that you will receive depends on whether or not you maintain the response and how you are able to tolerate ongoing therapy. There will be 4-8 weeks between each consolidation cycle depending on any side effects you may be having and your blood counts.

During consolidation cycles you will receive clofarabine on Days 1-3 by vein over 1-2 hours. You will receive cytarabine by injection under the skin over several seconds 2 times a day .

Induction and Consolidation Cycles:

On the days when you receive clofarabine and cytarabine (Days 1-5 during induction and Days 1-3 during consolidation), the clofarabine will be given about 3-6 hours before the cytarabine injections. You can be taught to give cytarabine injections to yourself. In this case, you can leave the clinic after receiving clofarabine. You will be required to record the injections of cytarabine in a diary unless you receive the treatments while you are in the hospital.

Study Visits:

On Day 1 of every cycle (+/- 7 days):

* You will have a physical exam, including measurements of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1-2 teaspoons) will be drawn for routine tests.

About 4 weeks after you started your first cycle, you may have a bone marrow aspirate to check the status of the disease. After that, you may have repeat bone marrow aspirates when the doctor thinks it is needed.

It is recommended that you stay in Houston for up to the first 4 weeks of treatment. After that, you will need to return to Houston before each induction cycle. If you continue with the consolidation you can receive these treatments by your local oncologist. However, you have to return to Houston at least every 3 months for your study visits.

Length of Study:

You may continue taking the study drugs for up to 15 cycles. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Clofarabine is FDA approved and commercially available for use in pediatric patients with acute lymphoblastic leukemia. Its use in adults and in patients with MDS is investigational.

Cytarabine is FDA approved and commercially available for use in patients with acute myeloid leukemia (AML).

Up to 80 patients will take part in this study. All be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years.
2. Diagnosis of MDS confirmed within 10 weeks prior to study entry according to World Health Organization (WHO) or French-American-British (FAB) criteria. Patients are either not eligible for or choose not to proceed with a stem cell transplant.
3. MDS classified as follows: refractory anemia with excess blasts (RAEB-1) (5%-9% BM blasts); RAEB-2 (10%-19% BM Blasts); chronic myelomonocytic leukemia (CMML) (5%-19% Bone Marrow (BM) blasts); RAEB-t (20%-29% BM blasts) AND/OR by International Prostate Symptom Score (IPSS): intermediate-2 and high risk patients.
4. No response, progression, or relapse (according to 2006 International Working Group (IWG) criteria; see section 8 for details) following at least 4 cycles of either azacitidine or decitabine, or following at least 2 cycles of SGI-110, which were completed within the last 2 years - AND/OR - intolerance to azacitidine, decitabine, or SGI-110 defined as drug-related >/= grade 3 hepatic or renal toxicity leading to treatment discontinuation during the preceding 2 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of </= 2.
6. Willing to adhere to and comply with all prohibitions and restrictions specified in the protocol.
7. Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
2. Active infection not adequately responding to appropriate antibiotics (i.e. ongoing temperatures of >/= 38 degree Celsius).
3. Total bilirubin >/= 1.5 mg/dL and not related to hemolysis or Gilbert's disease. Patients with total bilirubin >/= 1.5 mg/dL to 3 mg/dL are eligible if at least 75% of the bilirubin is indirect.
4. Alanine transaminase (ALT/SGPT) or aspartate transaminase (AST/SGOT) >/= 2.5 x the upper limit of normal.
5. Serum creatinine > 1.5 mg/dL.
6. Female patients who are pregnant or lactating.
7. Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices (IUD), double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study.
8. Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening.
9. Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy.
10. No prior treatment with cytarabine or clofarabine. Prior hydroxyurea for control of leukocytosis or use of hematopoietic growth factors (eg, G-CSF, Granulocyte-macrophage colony-stimulating factor (GM-CSF), procrit, aranesp, thrombopoietins) is allowed at any time prior to or during study if considered to be in the best interest of the patient.
11. Psychiatric illness or social situation that would limit the patient's ability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2017-01-29 (Actual); Study Completion 2017-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/2011 to 10/2015
Pre-assignment Details: Of the 81 participants registered, one participant was never treated with the study medication. All Participants were registered at The University of Texas MD Anderson Cancer Center.
Groups:
- Clofarabine + Cytarabine: Induction:
  Clofarabine 10 mg/m2 1-2 hours by vein daily for 5 days (days 1-5) Cytarabine 20 mg subcutaneously twice daily for 7 days (days 1-7)
  Consolidation:
  Clofarabine 10 mg/m2 1-2 hours by vein daily for 3 days (days 1-3) Cytarabine 20 mg subcutaneously twice daily for 5 days (days 1-5)
  Clofarabine: Induction:
  10 mg/m2 by vein over 1-2 hours daily for 5 days (days 1-5)
  Consolidation:
  10 mg/m2 by vein over 1-2 hours daily for 3 days (days 1-3)
  Cytarabine: Induction:
  20 mg subcutaneously twice daily for 7 days (days 1-7)
  Consolidation:
  20 mg subcutaneously twice daily for 5 days (days 1-5)
Period: Overall Study
Arm/Group | Clofarabine + Cytarabine
Started | 81
Completed | 80
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine + Cytarabine
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 65
Age, Continuous [Median (Full Range); unit: years] | 71 [30 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 72
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: Complete Response Criteria (CR must last for at least 4 weeks): Marrow: </= 5% myeloblasts with normal maturation of all cell lines; Persistent dysplasia noted; Blood: Hemoglobin (Hb) >/= 11 g/dL (untransfused, patient not on EPO); Neutrophils >/= 1x109/L (not on myeloid growth factor); Platelets >/= 100 * 109/L (not on thrombopoietic agent); No blasts. Bone marrow aspirate and/or biopsy at the end of course 1 (day 28 +/- 7 days). The method of Thall, Simon, and Estey used to monitor response.
Time Frame: 4 weeks after first cycle
Population: One of the eighty-one participants registered on the study were in evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine + Cytarabine
Number analyzed (Participants) | 80
Participants | 19

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time interval from study entry date to the date of death due to any cause, measured in days/months. Bayesian time-to-event model used to monitor overall survival.
Time Frame: 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Clofarabine + Cytarabine
Number analyzed (Participants) | 80
Months | 10.3 [0.5 to 62]

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent until 30 days after the last dose of drug. AE's can be collected for up to 15 cycles.
Arm/Group | Clofarabine + Cytarabine
All-Cause Mortality (participants affected / at risk) | 16/81
Serious Adverse Events (participants affected / at risk) | 57/81
Other Adverse Events (participants affected / at risk) | 46/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cytarabine (N=81)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal Ulcer (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated aspartate aminotransferase (AST) (Metabolism and nutrition disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Failure to Thrive (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever of Unknown Origin (General disorders) | 2 (3)
Hepatic Failure (Renal and urinary disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 7 (9)
Infusion Reaction (General disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 4 (7)
Lung Infection (Infections and infestations) | 22 (26)
Memory Impairment (Nervous system disorders) | 1 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1)
Neck Mass (General disorders) | 1 (1)
Neutropenic Fever (Infections and infestations) | 25 (33)
Pain (General disorders) | 1 (1)
Pericardial Tamponade (Cardiac disorders) | 1 (1)
Pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1)
Rectal Ulcer (Gastrointestinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 7 (7)
Severe Deconditioning (General disorders) | 1 (1)
Spinal Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncopal Event (Nervous system disorders) | 1 (1)
Worsening Sweet Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine + Cytarabine (N=81)
Constipation (Gastrointestinal disorders) | 13 (13)
Elevated Alanine Aminotransferase (Metabolism and nutrition disorders) | 17 (17)
Fatigue (General disorders) | 6 (6)
Headache (General disorders) | 12 (12)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 18 (18)
Nausea (Gastrointestinal disorders) | 15 (15)
Neutropenic Fever (Infections and infestations) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT01444742/Prot_SAP_000.pdf